CLINICAL TRIAL: NCT02664545
Title: A Prospective, Randomized, Controlled, Clinical Trial Evaluating the Non-Inferiority of Bridge-Enhanced Anterior Cruciate Ligament Repair (BEAR) to Anterior Cruciate Ligament Reconstruction With an Autologous Tendon Graft (ACLR)
Brief Title: Bridge-Enhanced ACL Repair vs ACL Reconstruction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Miach Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BEAR II TRIAL
Record Dates: First submitted 2016-01-20; First posted 2016-01-27 (Estimated); Results first posted 2024-01-10 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Anterior Cruciate Ligament Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Bridge-Enhanced ACL Repair (BEAR) (Experimental): The BEAR technique involves surgically placing a sponge (the BEAR scaffold) between the torn ends of the ACL, providing a scaffold for the ligament ends to grow into.
  Interventions: Device: BEAR Scaffold
- Tendon Graft (Active Comparator): ACL reconstruction is when a tendon graft (either two hamstring tendons from the back of the knee or bone-patellar tendon-bone graft from the front of the knee) is taken and used to replace the torn ACL.
  Interventions: Procedure: Tendon Graft

INTERVENTIONS:
Device: BEAR Scaffold — A sponge, or scaffold, which is surgically placed between the torn ligament ends and sutures are used to repair the torn anterior cruciate ligament.
  Arms: Bridge-Enhanced ACL Repair (BEAR)
Procedure: Tendon Graft — A graft of tendon (either two hamstring tendons from the back of the knee or bone-patellar tendon-bone graft from the front of the knee)
  Arms: Tendon Graft

SUMMARY:
The goal of this trial is to compare the efficacy of the Bridge-Enhanced Anterior Cruciate Ligament Repair (BEAR™) technique with the current method of treatment for anterior cruciate ligament (ACL) injuries, ACL reconstruction.

DETAILED DESCRIPTION:
Enrolled patients will be randomized to either the Bridge-Enhanced ACL Repair (BEAR) technique (new treatment) or an ACL reconstruction (current gold standard of treatment).

ELIGIBILITY:
Inclusion Criteria:

* Age: 14 to 35 years of age.
* Sex: Both male and female
* ACL: Complete tear
* Time from injury to surgery: ≤45 days
* MRI: ACL tissue present on pre-operative MRI - at least 50% of the ACL length must still be attached to the tibial plateau

Exclusion Criteria:

* Prior surgery on affected knee
* Prior joint infection on affected knee
* Regular use of tobacco or nicotine
* Use of corticosteroid within last 3 months
* History of chemotherapy treatment
* History of sickle cell disease
* History of anaphylaxis
* Any condition that could affect healing or infection risk (Diabetes, inflammatory arthritis, etc)
* Operative posterolateral corner injury (LCL complete tear, Biceps femoris tendon avulsion, tear of the arcuate ligament, tear of the popliteus ligament)
* Grade III medial collateral ligament injury
* Complete patellar dislocation
* Known allergy to bovine, beef or cow products

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2028-05-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Meng Yen, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Menghini D, Kaushal SG, Flannery SW, Ecklund K; BEAR Trial Team; Murray MM, Fleming BC, Kiapour AM, Proffen B, Sant N, Portilla G, Sanborn R, Freiberger C, Henderson R, Barnett S, Yen YM, Kramer DE, Micheli LJ. Changes in the Cross-Sectional Profile of Treated Anterior Cruciate Ligament Within 2 Years After Surgery. Orthop J Sports Med. 2022 Oct 14;10(10):23259671221127326. doi: 10.1177/23259671221127326. eCollection 2022 Oct. PMID 36263311
- [Derived] Sanborn RM, Badger GJ; BEAR Trial Team; Yen YM, Murray MM, Christino MA, Proffen B, Sant N, Barnett S, Fleming BC, Kramer DE, Micheli LJ. Psychological Readiness to Return to Sport at 6 Months Is Higher After Bridge-Enhanced ACL Restoration Than Autograft ACL Reconstruction: Results of a Prospective Randomized Clinical Trial. Orthop J Sports Med. 2022 Feb 9;10(2):23259671211070542. doi: 10.1177/23259671211070542. eCollection 2022 Feb. PMID 35155707
- [Derived] Barnett SC, Murray MM, Flannery SW; BEAR Trial Team; Menghini D, Fleming BC, Kiapour AM, Proffen B, Sant N, Portilla G, Sanborn R, Freiberger C, Henderson R, Ecklund K, Yen YM, Kramer D, Micheli L. ACL Size, but Not Signal Intensity, Is Influenced by Sex, Body Size, and Knee Anatomy. Orthop J Sports Med. 2021 Dec 17;9(12):23259671211063836. doi: 10.1177/23259671211063836. eCollection 2021 Dec. PMID 34988237
- [Derived] Barnett SC, Murray MM, Badger GJ; BEAR Trial Team; Yen YM, Kramer DE, Sanborn R, Kiapour A, Proffen B, Sant N, Fleming BC, Micheli LJ. Earlier Resolution of Symptoms and Return of Function After Bridge-Enhanced Anterior Cruciate Ligament Repair As Compared With Anterior Cruciate Ligament Reconstruction. Orthop J Sports Med. 2021 Nov 9;9(11):23259671211052530. doi: 10.1177/23259671211052530. eCollection 2021 Nov. PMID 34778483
- [Derived] Murray MM, Fleming BC, Badger GJ; BEAR Trial Team; Freiberger C, Henderson R, Barnett S, Kiapour A, Ecklund K, Proffen B, Sant N, Kramer DE, Micheli LJ, Yen YM. Bridge-Enhanced Anterior Cruciate Ligament Repair Is Not Inferior to Autograft Anterior Cruciate Ligament Reconstruction at 2 Years: Results of a Prospective Randomized Clinical Trial. Am J Sports Med. 2020 May;48(6):1305-1315. doi: 10.1177/0363546520913532. Epub 2020 Apr 16. PMID 32298131
- [Derived] Murray MM, Kiapour AM, Kalish LA, Ecklund K; BEAR Trial Team; Freiberger C, Henderson R, Kramer D, Micheli L, Yen YM, Fleming BC. Predictors of Healing Ligament Size and Magnetic Resonance Signal Intensity at 6 Months After Bridge-Enhanced Anterior Cruciate Ligament Repair. Am J Sports Med. 2019 May;47(6):1361-1369. doi: 10.1177/0363546519836087. Epub 2019 Apr 15. PMID 30986359

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol enrollment is the number of participants who had surgery, not the number of participants who were evaluated at baseline.
Period: Overall Study
Arm/Group | Bridge-Enhanced ACL Repair (BEAR) | Tendon Graft
Started | 65 | 35
Surgery | 65 | 35
Completed (Completed 2-year Primary Endpoint.) | 58 | 32
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Population: Baseline data analyzed for N=100 subjects screened.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bridge-Enhanced ACL Repair (BEAR) | Tendon Graft | Total
Number analyzed (Participants) | 65 | 35 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 43 | 21 | 64
  Between 18 and 65 years | 22 | 14 | 36
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.5 (5.2) | 19.8 (5.3) | 19.6 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 19 | 56
  Male | 28 | 16 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 64 | 35 | 99
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 56 | 27 | 83
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.7 (3.8) | 23.5 (4.6) | 24.3 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: International Knee Documentation Committee (IKDC) Subjective
Description: This is a survey taken by patients to report how their knee is working for them. The IKDC is graded by adding the results and converting the result to a number on a scale from 0 to 100. Scores range from 0 (lowest level of function and highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Time Frame: 2 years after surgery
Population: Multiple imputation used for missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bridge-Enhanced ACL Repair (BEAR) | Tendon Graft
Number analyzed (Participants) | 65 | 35
score on a scale | 88.6 (13.4) | 84.6 (13.3)

2. Primary Outcome: Instrumented Anteroposterior (AP) Laxity Testing
Description: This is a test of how stable the knee is.
  The anteroposterior (AP) knee laxity will be determined using a KT arthrometer at the 30lb (130N) setting on both knees of the subject at six months and 1, 2, 6 and 10 years after surgery (see Appendix C). Both sides will be covered with a sleeve so the licensed examiner cannot tell which is the operated knee or which procedure the patient had.
  Values for both knees will be recorded. For knee laxity, a difference of 2.0 mm in the side-to-side difference measurements at 2 years after surgery, the primary analysis, for the patients in the bridge-enhanced repair group vs. the ACL reconstruction group will be considered clinically significant.
Time Frame: 2 years after surgery
Population: Multiple imputation used for missing data.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bridge-Enhanced ACL Repair (BEAR) | Tendon Graft
Number analyzed (Participants) | 65 | 35
mm | 1.7 (3.2) | 1.8 (2.8)

3. Secondary Outcome: Prone Hamstring Strength at 6 Months
Description: Measured by a hand-held dynamometer on both the involved and contralateral knees, measured as injured knee as percent of non injured knee. The subject lies on their stomach and flexes their leg. The trainer puts the dynamometer near the ankle in the direction of extension. The subject pushes as hard as they can in the flexion direction, against the dynamometer. Ratio is calculated as the measurement of injured knee over measurement of non-injured knee.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of non injured knee
Arm/Group | Bridge-Enhanced ACL Repair (BEAR) | Tendon Graft
Number analyzed (Participants) | 65 | 35
percentage of non injured knee | 93.3 (23.6) | 59.1 (21.3)

4. Secondary Outcome: Return to Sport (RSI) Patient Reported Outcomes Score at 6 Months.
Description: This is a survey taken by patients to report how confident they are in returning to sports after the injury. The 12 questions on the ACL-RSI scale ask about the psychological effects of returning to sports. The ACL-RSI items are graded using an NRS (numeric rating scale) from 0 to 10. It has three domains: risk appraisal, confidence, and emotions. A total score between 0 and 100 is calculated by adding and averaging the scores for each item. Greater psychological preparation is indicated by higher scores.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bridge-Enhanced ACL Repair (BEAR) | Tendon Graft
Number analyzed (Participants) | 65 | 35
score on a scale | 71.5 (19.5) | 58.9 (24.1)

ADVERSE EVENTS:
Time Frame: Adverse Events measured at 2-year Primary Endpoint.
Arm/Group | Bridge-Enhanced ACL Repair (BEAR) | Tendon Graft
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/35
Serious Adverse Events (participants affected / at risk) | 16/65 | 5/35
Other Adverse Events (participants affected / at risk) | 34/65 | 11/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bridge-Enhanced ACL Repair (BEAR) (N=65) | Tendon Graft (N=35)
ACL Injury- No Surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ACL Second Surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
ACL Second Surgery with Meniscus (Musculoskeletal and connective tissue disorders) | 8 (8) | 1 (1)
Arthrofibrosis-Surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Knee Pain-Surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Meniscus-Surgery (Musculoskeletal and connective tissue disorders) | 7 (11) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bridge-Enhanced ACL Repair (BEAR) (N=65) | Tendon Graft (N=35)
ACL Injury- No Surgery (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Injury- Knee Other No Surgery (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)
Knee Pain- No Surgery (Musculoskeletal and connective tissue disorders) | 10 (11) | 4 (4)
Meniscus- No Surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (2)
Infection Knee-Superficial No Abx (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT02664545/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT02664545/SAP_001.pdf